CLINICAL TRIAL: NCT05705440
Title: A Phase 3b, Non-randomized, Open Label, Multi-country, Cohort Study to Describe the Safety of Study Participants Who Received RSVPreF3 Maternal Vaccination (Any Dose) or Controls From Previous RSV MAT Studies (RSV MAT-001, RSV MAT-004, RSV MAT-010, RSV MAT-011, RSV MAT-009, RSV MAT-012 and RSV MAT-039) During Any Pregnancy Conceived Post Vaccination/Control
Brief Title: A Follow-up Study to Describe the Safety of Study Participants Who Received RSVPreF3 Maternal Vaccination (Any Dose) or Controls From Previous RSV MAT Studies During Any Pregnancy Conceived Post Vaccination/Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 219510; 2022-003124-41 (EudraCT Number)
Record Dates: First submitted 2023-01-20; First posted 2023-01-30 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Pregnancy; RSVPreF3 vaccine; Safety; Follow-up study; Retrospective data; Prospective data
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- RSVPreF3 Group (Other): Participants received the RSVPreF3 vaccine during the prior RSV MAT studies (RSV MAT-001, RSV MAT-004, RSV MAT-011, RSV MAT-010, RSV MAT-009, RSV MAT-012 and RSV MAT-039) according to the vaccination schedule specific to each study.
  Interventions: Biological: RSVPreF3 vaccine
- Control Group (Other): Participants received any control (placebo, Tdap or influenza vaccine) during the prior RSV MAT studies (RSV MAT-001, RSV MAT-004, RSV MAT-011, RSV MAT-010, RSV MAT-009, RSV MAT-012 and RSV MAT-039) according to the vaccination schedule specific to each study.
  Interventions: Other: Control

INTERVENTIONS:
Biological: RSVPreF3 vaccine — No intervention is administered in this extension study. Participants received the RSVPreF3 vaccine during the prior RSV MAT studies (RSV MAT-001, RSV MAT-004, RSV MAT-010, RSV MAT-011, RSV MAT-009, RSV MAT-012 and RSV MAT-039) according to the vaccination schedule specific to each study. In all prior RSV MAT studies, participants received one dose of RSVPreF3 vaccine except in RSV MAT-011 study, where some participants received a second dose as well.
  Arms: RSVPreF3 Group
Other: Control — No intervention is administered in this extension study. Participants received any control (placebo, Tdap or influenza vaccine) during the prior RSV MAT studies (RSV MAT-001, RSV MAT-004, RSV MAT-010, RSV MAT-011, RSV MAT-009, RSV MAT-012 and RSV MAT-039) according to the vaccination schedule specific to each study. In all prior RSV MAT studies, participants received one dose of any control (placebo, Tdap or influenza vaccine).
  Arms: Control Group

SUMMARY:
The purpose of this follow-up study is to describe the safety in subsequent pregnancies in participants who were previously administered the RSVPreF3 maternal vaccine or control during any prior RSV MAT study.

The study participants enrolled in this follow-up study received RSVPreF3 maternal vaccination (any dose) or controls during the following prior RSV MAT studies: RSV MAT-001 (NCT03674177), RSV MAT-004 (NCT04126213), RSV MAT-010 (NCT05045144), RSV MAT-011 (NCT04138056), RSV MAT-009 (NCT04605159), RSV MAT-012 (NCT04980391) and RSV MAT-039 (NCT05169905).

No intervention will be administered in this study. The exposure was the intervention (either RSVPreF3 vaccine or control) received by the study participants in the above-mentioned prior RSV MAT studies.

ELIGIBILITY:
Inclusion Criteria:

Retrospective cohort

Adult/Adolescent Participant:

* Adult/Adolescent study participant from any of the prior RSV MAT studies who have either received RSV MAT vaccine or control (placebo, Tdap or influenza vaccine).
* Study participant:

  * who has reached 2 years+2 months post vaccine/control prior to/at enrolment or
  * who has not reached 2 years+2 months post vaccine/control prior to/at enrolment but is a Woman of Nonchildbearing Potential (WONCBP) at study enrolment, or recipient of bilateral tubal ligation prior to study enrolment.
* Study participant with any pregnancy conceived post vaccination/control, that has reached Day 42 post-delivery prior to/at enrollment.
* Provide signed and dated informed consent form.
* Be willing to comply with all study requirements and be available for the duration of the study.

Infant Participant:

* Participant live born as the result of a pregnancy followed in an adult/adolescent participant in this study.
* Signed and dated informed consent form obtained from the participant's parent(s)/LAR(s) prior to performance of any study-specific procedure.

Prospective cohort

Adult/Adolescent Participant:

* Adult/adolescent study participant from any of the prior RSV MAT studies who have either received RSV MAT vaccine or control (placebo, Tdap or influenza vaccine).
* Study participant:

  * who has not reached 2 years+2 months post vaccine/control prior to/at enrollment or
  * who has reached at least 2 years+2 months post vaccine/control but has an ongoing pregnancy (prior to Day 42 post-delivery) at enrollment. Participants who have reached 2 years post-vaccine/control before enrollment but are pregnant at enrollment will be enrolled and followed until Day 42 post-delivery for the pregnancy ongoing at enrollment.
* Female participants of childbearing potential.
* Provide signed and dated informed consent form.
* Be willing to comply with all study procedures and be available for the duration of the study.

Infant Participant:

* Participant live born as the result of a pregnancy followed in an adolescent/adult participant in this study.
* Participant's parent(s)/LAR(s), in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Signed and dated informed consent form obtained from the participant's parent(s)/LAR(s) prior to performance of any study-specific procedure.

Exclusion Criteria:

Adult/adolescent participant otherwise eligible for the prospective cohort:

• Woman of Nonchildbearing Potential (WONCBP) at study enrollment, or recipient of bilateral tubal ligation prior to study enrollment, if she has not conceived a pregnancy post-vaccine/control and does not plan to use any additional measures to attempt to conceive a pregnancy (e.g., sterilization reversal or IVF).

Infant participant:

• Child in care.

Ages: 9 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 3962 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Percentage of maternal participants reporting pregnancy outcomes from Day 1 up to Day 42 post-delivery of the first pregnancy conceived within 2 years post-vaccination | From Day 1 up to Day 42 post-delivery of the first pregnancy conceived within 2 years post-vaccination
Percentage of maternal participants reporting pregnancy related adverse events of special interest (AESIs) from Day 1 up to Day 42 post-delivery of the first pregnancy conceived within 2 years post-vaccination | From Day 1 up to Day 42 post-delivery of the first pregnancy conceived within 2 years post-vaccination
Percentage of infant participants reporting infant AESIs from birth up to Day 42 post-birth of the first pregnancy conceived within 2 years post-vaccination | From birth up to Day 42 post-birth of the first pregnancy conceived within 2 years post-vaccination

SECONDARY OUTCOMES:
Percentage of maternal participants reporting pregnancy outcomes from Day 1 up to Day 42 post-delivery of any pregnancy conceived within 2 years post-vaccination | From Day 1 up to Day 42 post-delivery of any pregnancy conceived within 2 years post-vaccination
Percentage of maternal participants reporting pregnancy related AESIs from Day 1 up to Day 42 post-delivery of any pregnancy conceived within 2 years post-vaccination | From Day 1 up to Day 42 post-delivery of any pregnancy conceived within 2 years post-vaccination
Percentage of infant participants reporting infant AESIs from birth up to Day 42 post-birth of any pregnancy conceived within 2 years post-vaccination | From birth up to Day 42 post-birth of any pregnancy conceived within 2 years post-vaccination
Percentage of maternal participants reporting selected pregnancy outcomes stratified by selected risk factors of those outcomes, from Day 1 up to Day 42 post-delivery of any pregnancy conceived within 2 years post-vaccination | From Day 1 up to Day 42 post-delivery of any pregnancy conceived within 2 years post-vaccination
Percentage of maternal participants reporting pregnancy related AESIs stratified by selected risk factors of those events, from Day 1 up to Day 42 post-delivery of any pregnancy conceived within 2 years post-vaccination | From Day 1 up to Day 42 post-delivery of any pregnancy conceived within 2 years post-vaccination
Percentage of infant participants reporting infant AESIs stratified by selected risk factors of those events, from birth up to Day 42 post-birth of any pregnancy conceived within 2 years post-vaccination | From birth up to Day 42 post-birth of any pregnancy conceived within 2 years post-vaccination
Percentage of maternal participants reporting selected pregnancy outcomes stratified by selected risk factors of those outcomes, from Day 1 up to Day 42 post-delivery of the first pregnancy conceived within 2 years post-vaccination | From Day 1 up to Day 42 post-delivery of the first pregnancy conceived within 2 years post-vaccination
Percentage of maternal participants reporting pregnancy related AESIs stratified by selected risk factors of those events, from Day 1 up to Day 42 post-delivery of the first pregnancy conceived within 2 years post-vaccination | From Day 1 up to Day 42 post-delivery of the first pregnancy conceived within 2 years post-vaccination
Percentage of infant participants reporting infant AESIs stratified by selected risk factors of those events, from birth up to Day 42 post-birth of the first pregnancy conceived within 2 years post-vaccination | From birth up to Day 42 post-birth of the first pregnancy conceived within 2 years post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (115):
- United States (24):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Burbank, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Saginaw, Michigan
  - GSK Investigational Site, Biloxi, Mississippi
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Englewood, Ohio
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Hendersonville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Keller, Texas
  - GSK Investigational Site, Lampasas, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, Weatherford, Texas
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Seattle, Washington
- Argentina (2):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Córdoba
- Australia (3):
  - GSK Investigational Site, South Brisbane, Queensland
  - GSK Investigational Site, Southport, Queensland
  - GSK Investigational Site, Clayton, Victoria
- Bangladesh (2):
  - GSK Investigational Site, Matlab
  - GSK Investigational Site, Sylhet
- Belgium (3):
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Sint-Niklaas
- Brazil (5):
  - GSK Investigational Site, Nova Iguaçu
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, RibeirAo PretoSP
  - GSK Investigational Site, Santa Maria
  - GSK Investigational Site, São José do Rio Preto
- Canada (12):
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, London-Ontario, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Joliette, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Colombia (4):
  - GSK Investigational Site, Barranquilla
  - GSK Investigational Site, Cali Colombia
  - GSK Investigational Site, Chía
  - GSK Investigational Site, Medellín
- GSK Investigational Site, Santo Domingo Este, Dominican Republic
- Finland (9):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- France (3):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Bron
  - GSK Investigational Site, Paris
- Germany (5):
  - GSK Investigational Site, Goch
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Hanover
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, Würzburg
- Honduras (2):
  - GSK Investigational Site, Comayagua
  - GSK Investigational Site, San Pedro Sula
- India (6):
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Mangalore
  - GSK Investigational Site, Mysore
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Vadu Budruk Pune
- Italy (4):
  - GSK Investigational Site, Bari
  - GSK Investigational Site, Messina
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Prato
- New Zealand (3):
  - GSK Investigational Site, Grafton Auckland
  - GSK Investigational Site, Papatoetoe Auckland
  - GSK Investigational Site, Wellington
- GSK Investigational Site, Panama City, Panama
- GSK Investigational Site, Manila, Philippines
- South Africa (4):
  - GSK Investigational Site, Johannesburg
  - GSK Investigational Site, Pretoria
  - GSK Investigational Site, Soshanguve
  - GSK Investigational Site, Soweto Gauteng
- South Korea (2):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Seoul
- Spain (14):
  - GSK Investigational Site, Aravaca
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Boadilla Del Monte Madrid
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Getafe
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, TorrejOn Ardoz Madrid
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Valladolid
- Taiwan (3):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/